CLINICAL TRIAL: NCT00627133
Title: A Pilot Study Examining the Efficacy of Keppra in Acute Alcohol Related Seizure Control in the Emergency Department Setting
Brief Title: Efficacy of Keppra in Acute Alcohol Related Seizure Control--A Pilot Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Keith Borg MD PhD, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K17644
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2008-02

CONDITIONS: Seizure, Alcohol Related
Keywords: Alcohol seizure
MeSH Terms: conditions — Alcohol Withdrawal Seizures | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: levetiracetam

INTERVENTIONS:
Drug: levetiracetam — 2 gram iv load, 500mg bid

SUMMARY:
Pilot study to evaluate efficacy of Keppra (levetiracetam) for seizure control in patients with alcohol related seizures.

ELIGIBILITY:
Inclusion Criteria:

* No trauma
* Not pregnant
* No other cause for seizure (hypoglycemia, CNS causes, trauma)
* Good family support
* Working telephone contact

Exclusion Criteria:

* Pregnancy
* Renal failure (creatine > 2mg/dl
* Fever or illness
* Hypotension
* Any trauma

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-02; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Decreased seizures | 1, 2, 4, 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States